CLINICAL TRIAL: NCT06831513
Title: A Pilot Study - to Observe the Effects of the Serkel Cranial Remolding Orthosis on Infants With Deformational Plagiocephaly, a Pre-market Fitting
Brief Title: Observe the Effects of the Serkel Cranial Remolding Orthosis on Infants With Deformational Plagiocephaly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Dara Spivey, Principle Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0287
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Plagiocephaly, Nonsynostotic
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic

STUDY DESIGN:
Intervention Model Description: Participants with deformational plagiocephaly, who qualify for cranial remolding treatment were fitted with a (new to US market) 3D printed cranial remolding orthosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Serkel 3D CRO Arm (Other): Once parents/caregivers decide and consent for their child to participate and be treated with the pre-market Serkel 3D CRO, infant's head will be scanned and CRO will be fabricated and fitted 2 weeks later. The orthosis is nearly identical to existing FDA approved devices.
  Interventions: Device: Serkel 3D CRO

INTERVENTIONS:
Device: Serkel 3D CRO — Serkel 3D CRO is intervention for those with deformational plagiocephaly and already qualified for a cranial remolding orthosis

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a specific brand of cranial remolding orthosis (a custom made helmet), which is new to the United States market

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and effectiveness of a specific brand of cranial remolding orthosis (a custom made helmet), which is new to the United States market. Serkel is an Australian company that specializes in the fabrication of 3D printed cranial remolding orthoses (CRO) to treat infants with deformational head shapes. Serkel has made over 600 helmets that have treated children with deformational head shapes in Australia, however it's specific helmet design is not FDA approved to provide treatment in the United States market. Serkel is seeking FDA approval of their brand of CRO by providing CRO's for pre market fitting. The study includes treatment for children who have been screened and diagnosed with a positional deformational head shape. Those who qualify for a FDA approved CRO treatment and were given the option to participate in the study. If they were interested, an inform consent provided and reviewed together. Cargivers then had the option to enroll. In total, 18 participants were enrolled. Fabrication scans were taken of the subjects head, and they returned 2 weeks later for fitting of the 3D printed cranial remolding orthosis, and seen for follow up every 2-4 weeks until treatment was complete (head shape corrected or participant outgrew CRO).

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 4-18 months at evaluation
* Participants with physician prescription of CRO treatment
* Participants with physician diagnosis of deformational plagiocephaly
* Participants who skulls measurements qualify them for standard CRO treatment (CVA measurement is greater than 6mm and Cephalic Index is greater than 92%)

Exclusion Criteria:

* Participants younger than 4 months at evaluation
* Participants older than 18 months at evaluation
* Participants without physician prescription for CRO treatment
* Participants without physician diagnosis of deformational plagiocephaly
* Participants whos skull measurements or asymmetries do not qualify them for standard CRO treatment

Ages: 4 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dara Spivey, MSOP, Principal Investigator — University of Texas Southwestern Prosthetics Orthotics
Locations (1):
- UTSouthwestern University - School of Health Professions, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 subjects consented but 1 screen failed and did not start treatment with the device. Therefore, only 18 considered enrolled and started treatment.
Period: Overall Study
Arm/Group | Serkel 3D CRO Arm
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Serkel 3D CRO Arm
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: weeks] | 30.4 [16 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 10
  Asian | 1
  Caucasian | 6
  African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Cranial Measurements as Measured by CVA
Description: Skull measurement are taken at every appointment the participant attends. At the end of treatment, the measurements will be compared to the participants starting measurements. Measurements can be taken by hand, using a tape measure and calipers. Or using an FDA approved scanner -- OMEGA Scanner 3D or Orthomerica STARscanner.
  * Cranial Vault Asymmetry (CVA) measures the difference between the lengths of two diagonals on the top of the skull. These diagonals are measured at a 30-degree angle from the midline. The CVA equation is: CVA = A - B, where A and B are the lengths of the longer and shorter diagonals, respectively. CVA is measured in millimeters.
Time Frame: Baseline, approximately 4-6 months
Measure: Mean (Full Range); unit: mm
Arm/Group | Serkel 3D CRO Arm
Number analyzed (Participants) | 18
mm
  Cranial Vault Asymmetry at start of treatment | 11.6 [3.5 to 18.4]
  Cranial Vault Asymmetry at end of treatment | 7.1 [.2 to 16.1]

2. Primary Outcome: Change in Cranial Measurements as Measured by Cephalic Index
Description: Skull measurement are taken at every appointment the participant attends. At the end of treatment, the measurements will be compared to the participants starting measurements. Measurements can be taken by hand, using a tape measure and calipers. Or using an FDA approved scanner -- OMEGA Scanner 3D or Orthomerica STARscanner.
  * The Cephalic Index (CI) is a measurement of head shape in infants, calculated by dividing head width by head length and multiplying by 100. A CI within the normal range (75-90%) indicates a typical head shape, while deviations, especially those leading to brachycephaly (CI > 90%) or dolichocephaly (CI < 76%), may be associated with developmental or medical concerns.
Time Frame: Baseline, approximately 4-6 months
Measure: Mean (Full Range); unit: percentage
Arm/Group | Serkel 3D CRO Arm
Number analyzed (Participants) | 18
percentage
  Cephalic Index at start of treatment | 89.8 [75.8 to 107.6]
  Cephalic Index at end of treatment | 86.8 [78.7 to 99.6]

ADVERSE EVENTS:
Time Frame: Adverse events data collection occurred every 2 or 3 weeks throughout the time the subject was enrolled in the trial. Subjects enrollment/treatment time varied based on age and severity of skull deformation. On average subjects were enrolled and receiving treatment for 22 weeks.
Arm/Group | Serkel 3D CRO Arm
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
A limitation was not having statistical analysis planned. Only a descriptive analysis was performed (start and completion of head shape measurements) and study was intended to collect de-identified data on a small sample size and never intended to publish.

The funding sponsor, Serkel, went bankrupt and the company dissolved shortly after trials were complete, the final de-indentified data was not shared with Serkel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT06831513/Prot_000.pdf